CLINICAL TRIAL: NCT05326165
Title: Preventing the Progression of Low Volume Swelling to Breast Cancer-related Lymphedema: a Pilot Study
Brief Title: Early Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Heinz Family Foundation (Unknown); Adele McKinnon Research Fund for Breast Cancer-Related Lymphedema (Unknown); Olayan-Xefos Family Fund for Breast Cancer Research (Unknown)
Responsible Party: Principal Investigator, Alphonse Taghian, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-600
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Breast Cancer Treatment Related Lymphedema
Keywords: Breast Cancer; Breast Cancer Treatment Related Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Breast Cancer Lymphedema | interventions — Gloves, Protective

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Compression therapy (Experimental): Participants will receive a ready to wear compression sleeve and glove with embedded sensor.
  Compression sleeve will be set to 20-30mm Hg pressure with instructions to wear for 12 hours a day for four consecutive weeks.
  Participants will also receive a journal to record usage and standard of care post-operative lymphedema monitoring and education and asked to fill out questionnaires.
  Interventions: Device: Juzo Compression Sleeve and Glove; Device: Compression Sleeve Sensor

INTERVENTIONS:
Device: Juzo Compression Sleeve and Glove — Elasticized garment sized for arm and hand to create pressure to reduce swelling
Device: Compression Sleeve Sensor — Small device embedded within compression sleeve garment collecting usage information

SUMMARY:
This research study is a Pilot Study examining the use of a compression sleeve with embedded sensor to prevent lymphedema.

DETAILED DESCRIPTION:
This is a single arm pilot study of a compression sleeve intervention for patients at high risk of breast cancer-related lymphedema (BCRL). The compression sleeve will also include a novel sensor to capture patient adherence to compression wear and pressure applied to the arm.

This research is being done because patients receiving lymph node surgery and lymph node radiation for breast cancer are at risk of lymphedema on the arm, trunk or breast/chest wall on the side of treatment. There is some evidence that compression sleeves may prevent progression of early swelling to lymphedema. This study is looking to determine if:

1. a compression garment worn for four weeks helps to prevent breast cancer-related lymphedema (BCRL) in those at high risk of BCRL
2. a sensor attached to the sleeve is accurately measuring time worn and pressure applied
3. participants are wearing the compression for the prescribed time, and if not, what are the barriers to wear
4. participants adhere to the study schedule for filling out patient surveys regarding symptoms and satisfaction with screening.

Findings from this study will apply to the development of a larger randomized controlled trial to examine if compression prevents progression to BCRL for patients with low volume swelling.

Study procedures include screening for eligibility, treatment including evaluations and follow up visits. Study treatment will last for four weeks with follow up at one, three, six, nine and 12 months.

It is expected that about 40 people will take part in this research study.

This study is receiving financial support from the Adele McKinnon Research Fund for Breast Cancer-Related Lymphedema (AG Taghian); the Olayan-Xefos Family Fund for Breast Cancer Research (AG Taghian), and the Heinz Family Foundation (AGTaghian).

Juzo Inc. is supporting this research study by providing compression garments and a Juzo pressure monitor. Impedimed Inc is supporting this study by providing a Sozo bioimpedance measurement device for research use.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be female, >/= 18 years, who underwent BC surgery for invasive or in-situ carcinoma with unilateral axillary lymph node dissection (ALND) (with or without contralateral prophylactic SLNB). Because of the extremely low incidence of BC in children and males, only female participants over the age of 18 will be included.
* Eligible participants will demonstrate low volume swelling (RVC 5-<10%) >/=12 weeks postoperatively
* Eligible participants will read and comprehend English, with the ability to understand and the willingness to sign a written consent document.
* Most patients treated for breast cancer will have undergone SLNB for axillary staging, and are therefore at lower risk for BCRL, compared to patients with ALND and/or regional lymph node radiation (RLNR). We have chosen to include only patients at high risk of BCRL, i.e., those who have undergone ALND, and we will not be including those who are at low BCRL risk, i.e., had only SLNB for axillary staging on the side of BC.

Exclusion Criteria:

* Participants who have bilateral BC (ie. contralateral staging SLNB or ALND) will not be eligible due to the need of a contralateral control arm for the RVC equation.
* Participants will not be eligible if they have been diagnosed and/or treated for BCRL.
* Participants will not be eligible if they have metastases that may cause BCRL. Participants with metastatic disease will be excluded.
* Participants with implanted cardiac devices and those who are pregnant will be excluded from the Sozo measurement component of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Arm Volume | 1, 3, 6, 9 and 12 months
  Primary objective is efficacy of compression intervention to change rate of progression from low volume swelling (LVS) (relative volume change (RVC) 5-<10%) to breast cancer-related lymphedema (BCRL) (RVC >/=10%). Measurement of effect of the compression intervention will be completed with arm volume measurements using perometry (infrared optical electronic scanner) .

SECONDARY OUTCOMES:
Sensor Accuracy | 4 Weeks
  Accuracy will be defined as sensor-detected wear within ±4.17% of true wear
Adherence rate to compression | 4 Weeks
  Percentage of participants who wear the garment for >/=50% of the instructed time (>/=6 of 12 instructed hours per calendar day), >57% of calendar days (>/=4 days per week),
Questionnaire Completion | 1, 3, 6, 9 and 12 months
  Percentage of participants who complete Breast Cancer and Lymphedema Symptom Experience Index and Functional Assessment of Cancer Therapy-- Breast Cancer questionnaires at each study visit per study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Alphonse G Taghian, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation